CLINICAL TRIAL: NCT02230904
Title: A Multicenter, Randomized, Double-blind, 2-way Cross-over Study to Compare the Adhesiveness of 2 Different Rotigotine Patch Formulations in Subjects With Parkinson's Disease
Brief Title: A Study to Compare the Adhesiveness of 2 Different Rotigotine Patches Used for the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Collaborators: Pharmaceutical Health Sciences (Unknown); Bracket Global (Unknown)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD0018; 2014-000932-41 (EudraCT Number)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson's Disease
Keywords: Rotigotine patch; Neupro; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm A-B (Experimental): 4 day treatment (Treatment A: Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1 followed by Treatment B: Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1)
  Interventions: Drug: Rotigotine (Test product PR 2.3.1); Drug: Rotigotine (Reference product PR 2.1.1)
- Treatment Arm B-A (Experimental): 4 day treatment (Treatment B: Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1 followed by Treatment A: Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1)
  Interventions: Drug: Rotigotine (Test product PR 2.3.1); Drug: Rotigotine (Reference product PR 2.1.1)

INTERVENTIONS:
Drug: Rotigotine (Test product PR 2.3.1) — * Pharmaceutical form: Transdermal patch
  * Concentration: 8 mg/24 hours
  * Route of administration: Transdermal
Drug: Rotigotine (Reference product PR 2.1.1) — * Pharmaceutical form: Transdermal patch
  * Concentration: 8 mg/24 hours
  * Route of administration: Transdermal
  Other Names: Neupro

SUMMARY:
The primary objective of the study is to compare the adhesiveness of 2 different patch formulations of Rotigotine using the largest patch size of 40 cm^2, under the assumption that both patch formulations show similar adhesiveness properties.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of idiopathic Parkinson's Disease
* Subject has been on continuous treatment with commercially available Rotigotine transdermal patches (Neupro®) for at least 3 months prior to enrollment
* Subject has been taking a stable Rotigotine dose including an 8 mg/24 hours (40 cm^2) patch for at least 2 weeks prior to enrollment

Exclusion Criteria:

* Subject has any medical or psychiatric condition which, in the opinion of the investigator, could jeopardize or would compromise the subject's well-being or ability to participate in this study
* Subject has a history of significant skin hypersensitivity to adhesives or other transdermal products or recently unsolved contact dermatitis
* Subject has a history or present condition of an atopic or eczematous Dermatitis, Psoriasis, or an active skin disease
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1) or Baseline (Visit 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (11):
- Germany (11):
  - 104, Alzenau in Unterfranken
  - 106, Aschaffenburg
  - 105, Berlin
  - 107, Böblingen
  - 101, Cologne
  - 111, Düsseldorf
  - 109, Erbach im Odenwald
  - 110, Essen
  - 102, Karlstadt am Main
  - 103, Stuttgart
  - 108, Würzburg

REFERENCES:
- [Derived] Elshoff JP, Bauer L, Goldammer N, Oortgiesen M, Pesch H, Timmermann L. Randomized, double-blind, crossover study of the adhesiveness of two formulations of rotigotine transdermal patch in patients with Parkinson's disease. Curr Med Res Opin. 2018 Jul;34(7):1293-1299. doi: 10.1080/03007995.2018.1430559. Epub 2018 Feb 20. PMID 29461870
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in September 2014 in Germany and concluded in December 2014.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Treatment Arm A-B: 4 day treatment (Treatment A for 2 days (Day 1 and Day 2): Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1 followed by Treatment B for 2 days (Day 3 and Day 4): Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1)
- Treatment Arm B-A: 4 day treatment (Treatment B for 2 days (Day 1 and Day 2): Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1 followed by Treatment A for 2 days (Day 3 and Day 4): Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1)
Period: Overall Study
Arm/Group | Treatment Arm A-B | Treatment Arm B-A
Started | 29 | 28
Completed | 29 | 27
Not Completed | 0 | 1
Not completed — Safety follow up could not take place | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set, consisting of all randomized subjects who entered the study and received at least 1 dose of study medication.
Arm/Group | Treatment Arm A-B | Treatment Arm B-A | Total Title
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.9) | 69.6 (9.5) | 68.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Adhesiveness Score of 2 Days of 24 Hours Patch Application as Rated by the Investigator (or Designee) Assessed According to the EMA Draft Guideline
Description: The assessment was performed according to the adhesion score adapted from the EMA draft guideline on quality of transdermal patches (EMA/CHMMP/QWP/911254/2011, 2012).
  * 0 = > 95 - 100 % of the patch area adheres
  * 1 = > 90 - 95 % of the patch adheres
  * 2 = > 85 - 90 % of the patch adheres
  * 3 = > 80 - 85 % of the patch adheres
  * 4 = > 75 - 80 % of the patch adheres
  * 5 = > 70 - 75 % of the patch adheres
  * 6 = ≥ 50 - 70 % of the patch adheres
  * 7 = < 50 % of the patch adheres
  * 8 = Patch completely detached
  The recorded scores 6, 7, and 8 were combined in order to create a cumulative group "less than or equal to 70 % adhered or patch detachment" which was regarded as significant patch adhesion failure in the draft EMA guideline.
  The average of patches 1 and 2 is presented by Treatment Arm below.
Time Frame: Patch adhesiveness was measured after 24 hours (±1 hour) after previous patch application on Day 2, 3, 4 and 5
Population: Per Protocol Set (PPS), which was defined as all subjects who had at least 1 patch adhesiveness assessment after 24 hours of patch application by the investigator (or designee) for both treatments.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment A: Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1 for 2 days (Day 1 and Day 2 for subjects in Treatment Sequence A-B and Day 3 and Day 4 for subjects in Treatment Sequence B-A).
- Treatment B: Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1 for 2 days (Day 1 and Day 2 for subjects in Treatment Sequence B-A and Day 3 and Day 4 for subjects in Treatment Sequence A-B).
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
units on a scale | 1.04 (1.33) | 2.15 (1.96)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; The change in average adhesiveness score was average score for Treatment B minus average score for Treatment A; Test type: Superiority or Other; Mean Difference (Final Values) = 1.115, Standard Deviation 1.635

2. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Investigator or Designee 24 Hours After Patch Application According to the EMA Draft Guideline for Patch 1
Description: The assessment was performed according to the adhesion score adapted from the EMA draft guideline on quality of transdermal patches (EMA/CHMMP/QWP/911254/2011, 2012).
  * 0 = >95 - 100 % of the patch area adheres
  * 1 = >90 - 95 % of the patch adheres
  * 2 = >85 - 90 % of the patch adheres
  * 3 = >80 - 85 % of the patch adheres
  * 4 = >75 - 80 % of the patch adheres
  * 5 = >70 - 75 % of the patch adheres
  * 6 = ≥50 - 70 % of the patch adheres
  * 7 = <50 % of the patch adheres
  * 8 = Patch completely detached
  The recorded scores 6, 7, and 8 were combined in order to create a cumulative group "less than or equal to 70 % adhered or patch detachment" which was regarded as significant patch adhesion failure in the draft EMA guideline.
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 2 and 4
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Groups:
- Treatment A: Rotigotine transdermal patch 8 mg/24 hours, test product PR 2.3.1
- Treatment B: Rotigotine transdermal patch 8 mg/24 hours reference product PR 2.1.1
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  > 95 % | 65.4 | 46.2
  > 90 % - 95 % | 11.5 | 17.3
  > 85 % - 90 % | 7.7 | 5.8
  > 80 % - 85 % | 3.8 | 9.6
  > 75 % - 80 % | 3.8 | 1.9
  > 70 % - 75 % | 0 | 1.9
  <= 70 % | 7.7 | 17.3
  Missing | 0 | 0

3. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Investigator 24 Hours After Patch Application According to the EMA Draft Guideline for Patch 2
Description: as for outcome 2
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 3 and 5
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  > 95 % | 71.2 | 36.5
  > 90 % - 95 % | 5.8 | 7.7
  > 85 % - 90 % | 3.8 | 9.6
  > 80 % - 85 % | 3.8 | 9.6
  > 75 % - 80 % | 3.8 | 9.6
  > 70 % - 75 % | 1.9 | 3.8
  <= 70 % | 9.6 | 23.1
  Missing | 0 | 0

4. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Investigator 24 Hours After Patch Application According to the FDA/Center for Drug Evaluation and Research (CDER) Score for Patch 1
Description: The assessment was performed according to the adhesion score adapted from the EMA draft guideline on quality of transdermal patches . Afterwards, EMA scores were translated into FDA/CDER scores:
  * 0 (>95-100% of patch adheres) >> 0 (FDA/CDER)
  * 1 (>90-95% of patch adheres) >> 0 (FDA/CDER)
  * 2 (>85-90% of patch adheres) >> 1 (FDA/CDER)
  * 3 (>80-85% of patch adheres) >> 1 (FDA/CDER)
  * 4 ( >75-80% of patch adheres) >> 1 (FDA/CDER)
  * 5 (>70-75% of patch adheres) >> 2 (FDA/CDER)
  * 6 (≥50-70% of patch adheres) >> 2 (FDA/CDER)
  * 7 (<50 % of patch adheres) >> 3 (FDA/CDER)
  * 8 (Patch completely detached) >> 4 (FDA/CDER)
  Due to a slight mismatch of limits between FDA scores 0 and 1 as compared to EMA scores 1 and 2, the theoretical value of exactly 90 % of adh. fell into score 1 with the FDA scoring. A similar limit mismatch occured at exactly 75 %. These mismatches may have resulted in a slightly worse estimation of the adh. with the FDA score as compared to previous adh. studies.
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 2 and 4
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  >= 90 % | 76.9 | 63.5
  75 % -< 90 % | 15.4 | 17.3
  50 % -< 75 % | 1.9 | 11.5
  < 50 % | 3.8 | 0
  Detached | 1.9 | 7.7
  Missing | 0 | 0

5. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Investigator 24 Hours After Patch Application According to the FDA/Center for Drug Evaluation and Research (CDER) Score for Patch 2
Description: as for outcome 4
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 3 and 5
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  >= 90 % | 76.9 | 44.2
  75 % -< 90 % | 11.5 | 28.8
  50 % -< 75 % | 3.8 | 17.3
  < 50 % | 7.7 | 3.8
  Detached | 0 | 5.8
  Missing | 0 | 0

6. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Subject 24 Hours After Patch Application for Patch 1
Description: The subject assessed the patch adhesiveness by using the following score:
  * 0 = Satisfied with adhesiveness
  * 1 = Moderately satisfied with adhesiveness
  * 2 = Moderately unsatisfied with adhesiveness
  * 3 = Unsatisfied with adhesiveness
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 2 and 4
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  0 = Satisfied with adhesiveness | 75.0 | 65.4
  1 = Moderately satisfied with adhesiveness | 17.3 | 13.5
  2 = Moderately unsatisfied with adhesiveness | 3.8 | 9.6
  3 = Unsatisfied with adhesiveness | 3.8 | 11.5

7. Secondary Outcome: Patch Adhesiveness Per Day as Rated by the Subject 24 Hours After Patch Application for Patch 2
Description: as for outcome 6
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 3 and 5
Population: as for outcome 1
Measure: Number; unit: percentage of patches
Units Other Than Participants: patches
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
Number analyzed (patches) | 52 | 52
percentage of patches
  0 = Satisfied with adhesiveness | 73.1 | 59.6
  1 = Moderately satisfied with adhesiveness | 15.4 | 26.9
  2 = Moderately unsatisfied with adhesiveness | 9.6 | 5.8
  3 = Unsatisfied with adhesiveness | 1.9 | 7.7

8. Secondary Outcome: Change in Average Patch Adhesiveness Score of 2 Days of 24 Hour Patch Application as Rated by the Investigator (or Designee), Assessed According to the FDA/Center for Drug Evaluation and Research (CDER) Score
Description: as for outcome 4
Time Frame: Patch adhesiveness was measured 24 hours (±1 hour) after previous patch application on Day 2, 3, 4 and 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 52 | 52
units on a scale | 0.40 (0.60) | 0.85 (1.03)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; The change in average adhesiveness score was average score for Treatment B minus average score for Treatment A; Test type: Superiority or Other; Mean Difference (Final Values) = 0.442, Standard Deviation 0.895

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events were collected from Visit 2 (Day 1) up to the Safety Follow-up Visit (Day 12).
Description: Adverse Events refer to the Safety Set, consisting of all randomized subjects who entered the study and received at least 1 dose of study medication.
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 7/57 | 1/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=57) | Treatment B (N=57)
Erythema (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days